CLINICAL TRIAL: NCT02796716
Title: Rapid Microbiological Diagnostics for MDRO Quantitative Identification and Resistance Phenotyping to Guide Antibiotic Selection in Wounded Warriors and Veterans - Task 3
Brief Title: Study of Accuracy of New Diagnostic Technology to Guide Rapid Antibiotic Treatment for Serious Infections
Status: Completed | Type: Observational
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Accelerate Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 14-1193
Record Dates: First submitted 2016-05-11; First posted 2016-06-13 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: INFECTIONS; Skin and Subcutaneous Tissue Bacterial Infections; Healthcare-associated Infection; Infection Due to Resistant Bacteria
Keywords: Wounded warriors; Battlefield infection; ESBL; MRSA; KPC
MeSH Terms: conditions — Infections; Cross Infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Testing on new technology called Accelerate ID/AST system

SUMMARY:
This research will test a new ultra-rapid technology (called ID/AST Accelerate system) that uses a digital microscope to identify bacteria based on their growth patterns. This method does not have to wait for bacteria to grow in a lab. The new method can identify the type of bacteria within 2 hours of receiving a specimen. The new method also shows the effect of selected antibiotics on the bacteria including multidrug resistant bacteria so that doctors know within 6 hours from specimen collection which antibiotic kills the bacteria.

To check the accuracy, speed and impact of the new method on antibiotic prescribing, investigators are proposing a study with two parts; The first part will test the accuracy and speed of the results obtained by the new method. The second part will test if having the results from the new method early would change the antibiotics prescribed to a patient in a simulation experiment. An independent infectious disease physician will be shown the results from the new method and asked if the results were accurate, would it change the antibiotic treatment for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Remnant sample from available from microbiology culture (respiratory, blood or tissue/skin) ordered as part of usual clinical care.

Exclusion Criteria:

* Insufficient sample volume available after sufficient aliquot removed for usual care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatient or outpatient with a sample being sent for microbiology culture (respiratory, blood or tissue/skin).
Sampling Method: Non-Probability Sample
Enrollment: 2102 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Difference in empiric antimicrobial use | 1.5 years
  Antibiotic use from the time of specimen collection until antibiotic susceptibility testing results are available to treating clinicians. Antibiotic use will be measured in days of therapy (DOT). DOT in usual care and simulated ID/AST Accelerate system will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Connie S Price, MD, Principal Investigator — Denver Health; Ivor S Douglas, MD, Principal Investigator — Denver Health
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No